CLINICAL TRIAL: NCT00238082
Title: The Effect of HFA-beclomethasone Dipropionate on Static Lung Volumes in COPD
Brief Title: The Effect of QVAR on Lung Functioning in Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-1277
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: COPD
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Emphysema; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic | interventions — Beclomethasone

INTERVENTIONS:
Drug: HFA-134A Beclomethasone DIpropionate (QVAR)

SUMMARY:
This is an investigator-sponsored research study to evaluate if treatment with HFA-134a beclomethasone (QVAR) has an effect on peripheral (or outer) airway inflammation and airway "remodeling" or scarring in subjects with COPD. Approximately 20 subjects with COPD will participate for approximately 7 weeks, with 10 receiving an active (BDP) inhaler with HFA-134a and 10 receiving a placebo.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis
* FEV1/FVC<70%
* FEV1 50-80% predicted
* Albuterol response of <12% and <200mL or methacholine PC20 > 8mg/mL
* RV > 120% predicted
* DLCO < 80%
* smokers and nonsmokers
* Lower age limit 45 years

Exclusion Criteria:

* Asthma
* Other chronic airway or parenchymal lung disease
* Other comorbid illness (including but not limited to DM, MI or CAD-related intervention in 6 months, neurologic disease, syncope)
* Use of any steroid (oral, IV, nasal, pulmonary) within 12 weeks
* Use of theophylline, leukotriene modifiers within 12 weeks
* Use of long-acting beta-agonists (formoterol, salmeterol) or anticholinergic (tiotropium)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1999-11 (Actual); Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Spirometric response (FEV1)
Lung volumes such as residual volume (RV), thoracic gas volume, total lung capacity (TLC) and the RV/TLC ratio

CONTACTS AND LOCATIONS:
Overall Officials: Richard Martin, MD, Principal Investigator — National Jewish Medical and Research Center faculty
Locations (1):
- National Jewish Medical and Research Center, Denver, Colorado, United States